CLINICAL TRIAL: NCT01101880
Title: Phase 2 Study Of Clofarabine With High Dose Cytarabine And G-CSF Priming In Adult Patients Less Than Age 65 With Newly Diagnosed Acute Myeloid Leukemia Or Advanced Myelodysplastic Syndrome and/or Advanced Myeloproliferative Neoplasm
Brief Title: Clofarabine, Cytarabine, and Filgrastim in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia, Advanced Myelodysplastic Syndrome, and/or Advanced Myeloproliferative Neoplasm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Pamela S Becker, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7144; NCI-2010-00282 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-09

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Refractory Anemia With Excess Blasts; Untreated Adult Acute Myeloid Leukemia; Myeloproliferative Neoplasm With 10% Blasts or Higher
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myelomonocytic, Chronic; Anemia, Refractory, with Excess of Blasts | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Clofarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemotherapy and colony stimulating factor) (Experimental): INDUCTION THERAPY: Patients receive filgrastim SC daily beginning the day prior to chemotherapy and continuing until blood counts recover. Patients receive clofarabine IV over 1 hour followed by cytarabine IV over 2 hours daily for 5 days.
  CONSOLIDATION THERAPY: Patients receive filgrastim SC daily for 5 days beginning the day prior to chemotherapy. Patients receive clofarabine IV over 1 hour followed by cytarabine IV over 2 hours daily for 4 days.
  Treatment with induction therapy may continue for up to 2 courses and treatment with consolidation therapy may continue for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: filgrastim; Drug: clofarabine; Drug: cytarabine

INTERVENTIONS:
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Drug: clofarabine — Given IV
  Other Names: CAFdA; Clofarex; Clolar
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside

SUMMARY:
This phase II trial is studying how well giving clofarabine and cytarabine together with filgrastim works in treating patients with newly diagnosed acute myeloid leukemia (AML), advanced myelodysplastic syndrome (MDS), and/or advanced myeloproliferative neoplasm. Drugs used in chemotherapy, such as clofarabine and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving the drugs in different doses may kill more cancer cells. Colony stimulating factors, such as filgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the complete remission (CR) rate of this regimen as compared with 7 + 3 standard induction with the 90 mg/m^2/dose of daunorubicin (historical control) in previously untreated patients with AML or advanced MDS or advanced myeloproliferative neoplasm less than age 65.

SECONDARY OBJECTIVES:

I. To determine the event free survival (EFS), overall survival (OS) and treatment related mortality of this regimen.

II. To assess the toxicity of this regimen in previously untreated patients. III. To determine whether 3 consolidation chemotherapy cycles consisting of G-CSF (filgrastim), clofarabine, and cytarabine (GCLAC) can be administered with prompt recovery of blood counts.

OUTLINE:

INDUCTION THERAPY: Patients receive filgrastim subcutaneously (SC) daily beginning the day prior to chemotherapy and continuing until blood counts recover. Patients receive clofarabine intravenously (IV) over 1 hour followed by cytarabine IV over 2 hours daily for 5 days.

CONSOLIDATION THERAPY: Patients receive filgrastim SC daily for 5 days beginning the day prior to chemotherapy. Patients receive clofarabine IV over 1 hour followed by cytarabine IV over 2 hours daily for 4 days.

Treatment with induction therapy may continue for up to 2 courses and treatment with consolidation therapy may continue for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia by World Health Organization (WHO) criteria (except acute promyelocytic leukemia), or myelodysplastic syndrome, RAEB-2 by WHO classification or advanced myeloproliferative neoplasm with >= 10% blasts in the bone marrow or peripheral blood, including chronic myelomonocytic leukemia (CMML)-2 by WHO classification
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 2
* Serum creatinine =< 1.0 mg/dL; if serum creatinine > 1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be > 60 mL/min/1.73 m^2 as calculated by the Modification of Diet in Renal Disease equation
* Serum bilirubin =< 1.5 x upper limit of normal (ULN) unless elevation is thought to be due to Gilbert's syndrome, hemolysis, or hepatic infiltration by the hematologic malignancy
* Aspartate transferase (AST)/alanine transferase (ALT) =< 2.5 x ULN unless elevation is thought to be due to hepatic infiltration by the hematologic malignancy
* Alkaline phosphatase =< 2.5 x ULN
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment
* Male and female patients must use an effective contraceptive method during the study and for a minimum of 90 days after study treatment

Exclusion Criteria:

* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol with the exception of intrathecal chemotherapy administered on days that are not concurrent with clofarabine and cytarabine
* No prior induction chemotherapy for AML; treatment with hydroxyurea is permitted; treatment with imides or hypomethylating agents for preceding hematological disorders is permitted
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment
* Patients with significant organ compromise due to systemic fungal, bacterial, viral, or other infection
* Pregnant or lactating patients
* Any significant concurrent illness, condition, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results
* Have had a diagnosis of another malignancy, unless the patient has been disease-free for at least 3 years following the completion of curative intent therapy including the following:

  * Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed
  * Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed
* Prior allogeneic stem cell transplant

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2013-06 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Becker, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - Stanford University, Stanford, California
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Becker PS, Medeiros BC, Stein AS, Othus M, Appelbaum FR, Forman SJ, Scott BL, Hendrie PC, Gardner KM, Pagel JM, Walter RB, Parks C, Wood BL, Abkowitz JL, Estey EH. G-CSF priming, clofarabine, and high dose cytarabine (GCLAC) for upfront treatment of acute myeloid leukemia, advanced myelodysplastic syndrome or advanced myeloproliferative neoplasm. Am J Hematol. 2015 Apr;90(4):295-300. doi: 10.1002/ajh.23927. Epub 2015 Jan 30. PMID 25545153

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Chemotherapy and Colony Stimulating Factor): INDUCTION THERAPY: Patients receive filgrastim SC daily beginning the day prior to chemotherapy and continuing until blood counts recover. Patients receive clofarabine IV over 1 hour followed by cytarabine IV over 2 hours daily for 5 days.
  CONSOLIDATION THERAPY: Patients receive filgrastim SC daily for 5 days beginning the day prior to chemotherapy. Patients receive clofarabine IV over 1 hour followed by cytarabine IV over 2 hours daily for 4 days.
  Treatment with induction therapy may continue for up to 2 courses and treatment with consolidation therapy may continue for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  filgrastim: Given SC
  clofarabine: Given IV
  cytarabine: Given IV
Period: Overall Study
Arm/Group | Treatment (Chemotherapy and Colony Stimulating Factor)
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy and Colony Stimulating Factor)
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 53 [22 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 27
Cytogenetic Risk Factor [Count of Participants; unit: Participants]
  Favorable | 4
  Intermediate | 32
  Unfavorable | 13
  Indeterminate | 1
Antecedent hematological disorder (AHD) [Count of Participants; unit: Participants] | 23
FLT3 ITD mutation status [Count of Participants; unit: Participants] — Number of participants with a FLT3 ITD mutation
  Participants | 10
WBC [Median (Full Range); unit: cells x 10^9/L] | 12 [0.8 to 761.3]
Peripheral Blast [Median (Full Range); unit: percent of white blood cells] | 16 [0 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Rates of Complete Remission and Complete Remission With Incomplete Recovery of Counts
Description: With 50 patients, the rates of these endpoints will be estimated with a standard error of 5 to 7 percentage points, depending on the observed rates. Complete remission is defined as less than 5% blast cells present in the bone marrow and count recovery (absolute neutrophil count greater than 1000/microL and platelet count greater than 100,000/microL). Complete remission with incomplete recovery of counts is defined as less than 5% blast cells present in the bone marrow without compete count recovery (absolute neutrophil count less than 1000/microL and platelet count less than 100,000/microL).
Time Frame: Up to 5 years
Population: CR achieved with no AHD only applies to those who did not have AHD.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy and Colony Stimulating Factor)
Number analyzed (Participants) | 50
Participants
  CR achieved | 38
  CR achieved with first course of induction | 33
  CR + CRp achieved | 41
  CR achieved with no AHD: number analyzed (Participants) | 27
  CR achieved with no AHD | 23
  CR achieved with AHD: number analyzed (Participants) | 23
  CR achieved with AHD | 15
  CR + CRp achieved with AHD: number analyzed (Participants) | 23
  CR + CRp achieved with AHD | 18
  CR achieved with FLT3 positive: number analyzed (Participants) | 10
  CR achieved with FLT3 positive | 7
  CR achieved with favorable risk cytogenetics: number analyzed (Participants) | 4
  CR achieved with favorable risk cytogenetics | 4
  CR achieved with intermediate risk cytogenetics: number analyzed (Participants) | 32
  CR achieved with intermediate risk cytogenetics | 26
  CR + CRp achieved with intermediate risk cyto.: number analyzed (Participants) | 32
  CR + CRp achieved with intermediate risk cyto. | 27
  CR achieved with unfavorable risk cytogenetics: number analyzed (Participants) | 13
  CR achieved with unfavorable risk cytogenetics | 8
  CR + CRp achieved with unfavorable risk cyto.: number analyzed (Participants) | 13
  CR + CRp achieved with unfavorable risk cyto. | 10

2. Primary Outcome: Duration of Remission
Description: With 50 patients, the rates of these endpoints will be estimated with a standard error of 5 to 7 percentage points, depending on the observed rates. Remission is defined as less than 5% blasts in the bone marrow, no appearance of blasts in the peripheral blood, and no extramedullary disease (appearance of leukemic cells in other tissues).
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: weeks
Arm/Group | Treatment (Chemotherapy and Colony Stimulating Factor)
Number analyzed (Participants) | 9
weeks | 7 [4 to 84]

3. Primary Outcome: Time to Progression
Description: With 50 patients, the rates of these endpoints will be estimated with a standard error of 5 to 7 percentage points, depending on the observed rates.
Time Frame: Up to 5 years
Measure: Median (Full Range); unit: weeks
Arm/Group | Treatment (Chemotherapy and Colony Stimulating Factor)
Number analyzed (Participants) | 9
weeks | 7 [4 to 84]

4. Primary Outcome: Event Free Survival
Description: Number of patients in remission at a median follow up of 15 months.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy and Colony Stimulating Factor)
Number analyzed (Participants) | 50
Participants | 21

5. Primary Outcome: Treatment-related Mortality (TRM)
Description: Treatment-related mortality (TRM) data was not collected.
Time Frame: Up to 5 years
Population: Treatment-related mortality (TRM) data was not collected.
Arm/Group | Treatment (Chemotherapy and Colony Stimulating Factor)
Number analyzed (Participants) | 0

6. Primary Outcome: Overall Survival
Description: as for outcome 3
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Chemotherapy and Colony Stimulating Factor)
Number analyzed (Participants) | 50
months | 24.3 [15 to 60]

ADVERSE EVENTS:
Description: Other [Not including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Treatment (Chemotherapy and Colony Stimulating Factor)
Serious Adverse Events (participants affected / at risk) | 50/50
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy and Colony Stimulating Factor) (N=50)
infection (Infections and infestations) | 50 (95)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 31 (31)
Liver enzymes (Hepatobiliary disorders) | 20 (20)
Gastrointestinal (Gastrointestinal disorders) | 10 (10)
Metabolic (Metabolism and nutrition disorders) | 10 (10)
Dermatologic (Skin and subcutaneous tissue disorders) | 10 (10)
Neurologic (Nervous system disorders) | 6 (6)
Coagulation (Blood and lymphatic system disorders) | 4 (4)
Cardiovascular (Cardiac disorders) | 2 (2)
Ocular (Eye disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Hepatobiliary (Hepatobiliary disorders) | 1 (1)
Urinary (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No